CLINICAL TRIAL: NCT00289575
Title: Evaluation of Safety and Performance of Macroporous Biphasic Calcium Phosphate Granules Combined With Cellulosic-Derived Gel, in Filling Bones Gap After Aseptic Osteonecrosis Biopsy of Femur Head.
Brief Title: MBCP Safety and Performance in the Osteonecrosis of Femur Head
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomatlante (Industry)
Collaborators: CIC Bordeaux (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Osteonecrosis
Keywords: Femur head aseptic osteonecrosis; Bone reconstruction; Macroporous biphasic calcium phosphate granules
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MBCP

SUMMARY:
The aim of this pilot study is to evaluate MBCP performance in bone regeneration after osteonecrosis biopsy of the femur head. This technic may prevent the neck of the femur bone weakness following the healthy area drilling, thanks to a bone reconstruction at the expense of the biomaterial.

DETAILED DESCRIPTION:
Twelve patients will be enrolled in this study and evaluation of infection and inflammation of the drilled area, pain and hip function will be assessed during a one year follow up. Bone reconstruction will be evaluated with scanner and radiography.

ELIGIBILITY:
Inclusion Criteria:

* femur head osteonecrosis (1 to 2 level in ARCO scale)
* signed informed consent

Exclusion Criteria:

* primary bone infection
* femur head sphericity loss
* cancer, diabetes, tuberculosis previous history
* HIV, Hepatitis B, Hepatitis C infection
* drepanocytosis
* current corticotherapy
* current immunosuppressive therapy
* innate or acquired immune deficience
* pregnancy or lack of efficient contraception
* current participation in an other study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-02; Study Completion 2008-02

PRIMARY OUTCOMES:
Infection and inflammation of the drilled area (blood and clinical assessment).
Adverse events.

SECONDARY OUTCOMES:
Pain (Analogic Visual Scale)
Hip function
Bone reconstruction evaluation through scanner and radiography

CONTACTS AND LOCATIONS:
Overall Officials: Thierry FABRE, Pr, Principal Investigator — University Hospital, Bordeaux; Jacques DEMOTES-MAINARD, Pr, Study Chair — Clinical Research Center INSERM/Bordeaux University Hospital
Locations (1):
- Service de chirurgie orthopédique et traumatologique- Hôpital Pellegrin, Bordeaux, France